CLINICAL TRIAL: NCT00358865
Title: Checking the Usability of Video Projected Virtual Reality Sytem in Children With Acquired Brain Injury
Brief Title: Checking the Usability of a Virtual Reality System in Children With Brain Injury
Status: Completed | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Other Study IDs: SHEBA-05-3847-AB-CTIL
Record Dates: First submitted 2006-07-31; First posted 2006-08-01 (Estimated); Last update posted 2008-05-07 (Estimated); Status verified 2008-04

CONDITIONS: Acquired Brain Injury
Keywords: Virtual Reality; ABI; Projected system
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to check the usability of Virtual Reality (VR) Video Capture Projected System in children with acquired brain injury(ABI)and comparing their performance to the performance of normally developing children. The trial shall include 15 subjects in each group, aged 6-12 years old. ABI subjects are hospitalized at the hospital's Pediatric Rehabilitation Department Each subject will experience 3 different virtual environments. The subjects in the trial group will practice 3 experiences (3 times in 3 different days) during a period of a week to 10 days, to check the practice effect.In addition, all subjects will be tested in three tests: "PEDI" - to evaluate the functional abilities of daily living (dressing, eating...),The "Melbourne Assessment" - to evaluate functional movements of upper extremities, and the TEA-ch - to evaluate different attention abilities. Performance correlations will be tested between these tests and the performance in the VR first experience.

DETAILED DESCRIPTION:
The purpose of this study is to check the usability of Virtual Reality (VR) Video Capture Projected System in children with acquired brain injury(ABI) comparing their performance with the performance of normally developing children, matched by age, gender,sector and parents' education. subjects' age: 6 - 12 years old. The trial shall include 15 subjects in each group. ABI subjects are hospitalized at Sheba Hospital's Pediatric Rehabilitation Department.

Each subject will experience 3 different virtual environments. The subjects in the trial group will practice 3 experiences (3 times in 3 different days) during a period of a week to 10 days, to check the practice effect. In addition, all subjects will be tested in three tests: "PEDI" - to evaluate the functional abilities of daily living (dressing, eating...),The "Melbourne Assessment" - to evaluate functional movements of upper extremities, and the TEA-ch - to evaluate difference attention abilities.

Correlations between those tests to the performance in the VR experiences will be checked with Pearson's statistical correlation tests. The differences between the trial group (ABI children) and the control group will be checked with Independent t-tests.

ELIGIBILITY:
Inclusion Criteria:(trial group)

* acquired brain injury as a result of brain tumor excision intervention, traumatic brain injury, infection, vascular disorders, metabolic disorders or anoxia.
* ability to move at least one of the upper extremities against gravity in a partial range of motion (MMT: -3)

Exclusion Criteria: (trial group)

* Significant visual limitations
* Premorbid, progressive mental disorder or neurological injury
* Premorbid learning disability

Inclusion Criteria (control group):

* healthy subjects

Exclusion Criteria (control group):

* developmental disorders
* significant medical problems
* neurological disorders

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study sample consisted of 33 children, and was divided into study and control groups: 16 children with ABI from the Pediatric Rehabilitation department at the Sheba Medical Center, Tel Hashomer in the study group (mean age = 7.91, S.D. = 1.43, range from 6 to 11.4 years old), and 17 healthy participants in the control group (mean age = 7.94, S.D. = 1.57, range from 6 - 11.33 years).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2005-12; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: amichay brezner, PhD, Principal Investigator — Sheba Medical Center; Tamar Weiss, prof., Study Director — Haifa university, OT Department; Brat Orit, PhD, Study Director — Tel Aviv University, OT Department
Locations (1):
- Tel Hashomer (THS) - Pediatric Rehabilitation Department, Ramat Gan, Israel